CLINICAL TRIAL: NCT05690438
Title: Prediction of the Post-intensive Care Syndrome
Acronym: PREPICS
Status: Completed | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anna Milton, Principal investigator, Region Stockholm
Other Study IDs: Dnr KS K2022-4466
Record Dates: First submitted 2022-12-01; First posted 2023-01-19 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Critical Care
Keywords: Post-intensive care syndrome; Depression; Anxiety; Post-traumatic stress; Physical disability; Pain; Frailty; Resilience
MeSH Terms: conditions — postintensive care syndrome; Depression; Anxiety Disorders; Pain; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to assess whether a screening of patients at discharge from the intensive care unit (ICU) can predict psychological and physical problems three months later.

The main questions to answer are:

1. Can the screening method at ICU discharge predict psychological symptoms three months after ICU stay?
2. Can the screening method at ICU discharge predict new-onset physical disability three months after ICU stay?
3. Does pain, resilience (the individuals' ability to handle distress) and frailty affect the risk of developing psychological and physical problems three months after ICU stay? All adult patients with an ICU stay 12 hours or longer will be assessed for inclusion in the study. Three months after discharge from the ICU included patients will be asked to digitally answer a set of questionnaires, rating symptoms of depression, anxiety, post-traumatic stress and ability to perform activities of daily living. Patients will also be asked to state their health-related quality of life and on-going pain, how the pain affects their everyday life and the ability to endure difficult situations.

DETAILED DESCRIPTION:
Firstly, the investigators hypothesize that two novel screening instruments, developed by the research group, for identification of intensive care unit (ICU) survivors with elevated risk for psychological and physical morbidity have high external validity. Secondly, the investigators hypothesize that frailty, pain and resilience will affect the probability of developing post-intensive care syndrome (PICS) three months post-ICU.

The specific objectives with the project are:

1. To assess the predictive value and hence the validity of a screening instrument assessing the risk for

   1. psychological problems (study I)
   2. new-onset physical disability (study II) three months post-ICU
2. To evaluate if pain, frailty and resilience, i.e the individual's ability to handle distress, affect the development of PICS three months post-ICU (study III)
3. To assess individual daily wellbeing with a digital diary (study IV)

Studies I-III are observational cohort studies including 800 adult patients admitted to the ICU for a minimum of 12 hours. Consecutively discharged ICU patients will be assessed with the PROGRESS-ICU screening instruments, generating an individual risk in percentage for a) psychological problems and b) new-onset physical disability three months post-ICU. The instruments consists of questions regarding depressive symptoms, traumatic memories from the ICU stay, social support and age and an evaluation of the patient´s physical status at ICU discharge, assessed with the first five items of the Chelsea Critical Care Physical Assessment Tool, CPAx. Patients will also be asked to state their level of pain at discharge with a numeric rating scale (NRS). Basic demographics will be collected from the patient data management system, such as sex, admission diagnosis, severity of illness, ICU length of stay and duration of mechanical ventilation. Patients or next of kin will also be asked to state the patients' level of independence in performing ten different ADLs two weeks prior to hospitalisation, assessed with the Barthel Index (BI). Frailty will be assessed with the Clinical Frailty Scale (CFS).

Three months after ICU discharge, patients will be asked to digitally, or on paper by regular mail, fill out validated questionnaires assessing level of symptoms of depression, anxiety (Hospital Anxiety and Depression Scale (HADS)) and post-traumatic stress (Post-Traumatic Stress Symptom 14-question inventory (PTSS-14)). New-onset physical disability will be assessed with the Barthel index (BI), a questionnaire assessing the level of independency in performing activities of daily living. In accordance with the cut-offs recommended in the literature, and level used for caseness in the studies developing the screening instruments, a HADS subscale score ≥11 and a PTSS-14 part B score >45 will define clinically substantial psychological symptoms 24,25. A BI score reduction of ≥10 compared to baseline will define substantial new-onset physical disability and is close to the minimum clinically important difference suggested for the BI. At the three months follow-up patients will also be assessed regarding pain with the NRS and resilience with the modified version of the validated questionnaire Psychological Inflexibility in Pain Scale (PIPS), addressing the tendency to avoid situations that could imply pain or other discomforts. Self-efficay will also be assessed, i.e. the belief in one's ability to handle distress as a measure of resilience with the General self-efficacy scale. Health-related quality of life will be assessed with the RAND-36. The investigators also plan to perform psychometric testing of the questionnaires used and validate them in Swedish for the relevant population.

In a subgroup of patients (n=15) daily wellbeing will be evaluated with a digital diary where patients will be asked to answer short questions regarding their present mood twice a day for a total of 30 days (14 days in a row, with a pause for 4 weeks and a new 14-day period of digital diary questions). The questions will be available to patients via an application in a smartphone/tablet, reminding them to answer the questions twice a day through a message/push notification. This will render multiple data points for each individual enabling analyses of the development over time as well as individual variations. Fifteen participants are deemed sufficient for a first analysis of aggregated individual data. This type of data is also an important step towards the next phase, to develop tailored interventions matching the specific needs of the individual ICU survivor.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥18 years old, with an ICU stay ≥12 hours, surviving to ICU discharge.

Exclusion Criteria:

* No home address
* Dementia or other major cognitive dysfunction
* Unsufficient knowledge of the Swedish language for answering follow-up questionnaires
* Two or more limitations of treatment or moribund patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General adult ICU population, all admitted patients will be consecutively screened for inclusion.
Sampling Method: Probability Sample
Enrollment: 773 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Predictive accuracy of a psychological screening method | Outcome measured three months after ICU discharge
  Validation of a previously developed screening method for psychological problems three months post-ICU
Predictive accuracy of a physical screening method | Outcome measured three months after ICU discharge
  Validation of a previously developed screening method for physical problems three months post-ICU
Frailty (assessed with the clinical frailty scale) and psychological outcome after ICU stay, assessed with the Hospital Anxiety and Depression Scale. | Outcome measured three months after ICU discharge
  Assessment of associations between frailty (assessed with the clinical frailty scale) and the development of symptoms of depression and anxiety post-ICU.
Frailty (assessed with the clinical frailty scale) and psychological outcome after ICU stay, assessed with the Post-Traumatic Stress 14-Question Inventory. | Outcome measured three months after ICU discharge
  Assessment of associations between frailty (assessed with the clinical frailty scale) and the development of the post-traumatic stress symptoms.
Frailty (assessed with the clinical frailty scale) and physical outcome after ICU stay, assessed with the Barthel Index. | Outcome measured three months after ICU discharge
  Assessment of associations between frailty (assessed with the clinical frailty scale) and the development of the post-intensive care syndrome physical problems.
Pain (assessed with the numeric rating scale, NRS) and physical outcome after ICU stay, assessed with the Barthel Index. | Outcome measured three months after ICU discharge
  Assessment of associations between pain and the development of the post-intensive care syndrome physical aspects.
Pain (assessed with the numeric rating scale, NRS) and psychological outcome after ICU stay, assessed with the Post-Traumatic Stress 14-Question Inventory. | Outcome measured three months after ICU discharge
  Assessment of associations between pain and the development of symptoms of post-traumatic stress post-ICU.
Pain (assessed with the numeric rating scale, NRS) and psychological outcome after ICU stay, assessed with the Hospital Anxiety and Depression Scale. | Outcome measured three months after ICU discharge
  Assessment of associations between pain and the development of symptoms of depression and anxiety post-ICU.
Resilience (assessed with the general self-efficacy scale, the pain catastrophizing scale and the psychological inflexibility in pain scale) and physical outcome after ICU stay (assessed with the Barthel Index). | Outcome measured three months after ICU discharge
  Assessment of associations between resilience and the development of the post-intensive care syndrome physical problems.
Resilience (assessed with the general self-efficacy scale, the pain catastrophizing scale and the psychological inflexibility in pain scale) and psychological outcome after ICU stay, assessed with the Hospital Anxiety and Depression Scale. | Outcome measured three months after ICU discharge
  Assessment of associations between resilience and the development of symptoms of depression and anxiety post-ICU.
Resilience (assessed with the general self-efficacy scale, the pain catastrophizing scale and the psychological inflexibility in pain scale) and psychological outcome after ICU stay | Outcome measured three months after ICU discharge
  Assessment of associations between resilience and the development of symptoms of post-traumatic stress post-ICU.
Feasibility of a daily digital diary in ICU survivors | Diary questions during 14 + 14 days after ICU discharge, questionnaire at termination of the diary.
  Feasibility of a digital diary post-ICU assessed with a patient questionnaire at the end of the diary period and number of and reason for drop out.
Daily variations of well-being in ICU survivors | Digital diary questions during 14 + 14 days after ICU discharge, with follow-up questionnaires three months post-ICU
  Digital diary with questions related to well-being for individual ICU survivors for a total of 30 days (14 + 14 days with a 4-week pause in between) post-ICU discharge.
With-in person associations between cognitive-affective state and daily well-being in ICU survivors | Digital diary questions during 14 + 14 days after ICU discharge, with follow-up questionnaires three months post-ICU
  Daily diary questions on mood and cognitive state and associations with daily well-being questions (sleep, tiredness, stress) post-ICU discharge.
Associations between high daily patterns of cognitive-affective state between individuals and psychological recovery | Digital diary questions during 14 + 14 days after ICU discharge, with follow-up questionnaires three months post-ICU
  Daily diary questions on mood and cognitive state and associations with symptoms of depression, anxiety and post-traumatic stress post-ICU discharge.

SECONDARY OUTCOMES:
Health-related quality of life in patients with psychological and/or physical problems post-ICU | Inclusion during one year, follow-up three months post-ICU discharge
  Health-related quality of life assessed with the RAND-36
Health-related quality of life in patients with pain post-ICU | Inclusion during one year, follow-up three months post-ICU discharge
  HRQL assessed with the RAND-36
Health-related quality of life and associations with pre-ICU frailty assessed with the Clinical Frailty Scale. | Inclusion during one year, follow-up three months post-ICU discharge
  HRQL assessed with the RAND-36, frailty with the clinical frailty scale.
Health-related quality of life and associations with resilience | Inclusion during one year, follow-up three months post-ICU discharge
  HRQL assessed with the RAND-36
Validation of questionnaires in a Swedish ICU population and psychometric testing | One year
  Used questionnaires will be validated in a Swedish ICU population and psychometric testing will be performed.
Clinical frailty, assessed with the Clinical Frailty Scale, and ICU length-of-stay | Outcome measured at discharge from the ICU
  Clinical frailty and associations with ICU length-of-stay
Clinical frailty, assessed with the Clinical Frailty Scale, and duration of mechanical ventilation in ICU | Outcome measured at discharge from the ICU
  Clinical frailty and associations with duration of mechanical ventilation in ICU
Clinical frailty, assessed with the Clinical Frailty Scale, and symptoms of psychological problems post-ICU assessed with the Hospital Anxiety and Depression Scale. | Outcome measured three months after discharge from the ICU
  Clinical frailty and associations with symptoms of depression and anxiety three months post-ICU
Clinical frailty, assessed with the Clinical Frailty Scale, and symptoms of post-traumatic stress post-ICU assessed with the Post-Traumatic Stress Symptom 14-Question Inventory. | Outcome measured three months after discharge from the ICU
  Clinical frailty and associations with symptoms of post-traumatic stress three months post-ICU
Clinical frailty, assessed with the Clinical Frailty Scale, and physical performance at ICU discharge assessed with the Chelsea Critical care physical assessment tool | Outcome measured at discharge from the ICU
  Clinical frailty and associations with physical status at ICU discharge
Clinical frailty, assessed with the Clinical Frailty Scale, and ICU mortality. | Outcome measured at discharge from the ICU
  Clinical frailty and associations with ICU mortality
Clinical frailty, assessed with the Clinical Frailty Scale, and three-month physical function assessed with the Barthel Index. | Outcome measured three months after discharge from the ICU
  Clinical frailty and associations with post-ICU physical functioning.

OTHER OUTCOMES:
Physical function at ICU discharge and mortality | Three months
  Physical function at discharge from the ICU, assessed with the first five items of the Chelsea Critical Care Physical Assessment Tool (CPAx) and associations with mortality within three months post-ICU

CONTACTS AND LOCATIONS:
Overall Officials: Anna Milton, Principal Investigator — Karolinska Institutet/Karolinska University Hospital
Locations (4):
- Sweden (4):
  - Karolinska University Hospital, Stockholm
  - Capio S:t Göran's Hospital, Stockholm
  - Danderyd's Hospital, Stockholm
  - Södersjukhuset, Stockholm